CLINICAL TRIAL: NCT05231655
Title: Ex Vivo Multi Drug Screening of Solid Tumours to Determine Personalised Therapy Efficacy and Resistance
Brief Title: Ex VIvo DEtermiNed Cancer Therapy
Acronym: EVIDENT
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH20854
Record Dates: First submitted 2022-01-31; First posted 2022-02-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer; Kidney Cancer; Melanoma; Sarcoma; Glioblastoma; Head and Neck Cancer
Keywords: Personalized medicine; Ex vivo drug screen; Image based analysis
MeSH Terms: conditions — Urinary Bladder Neoplasms; Kidney Neoplasms; Melanoma; Sarcoma; Glioblastoma; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be retained for the duration of the study where surplus tissue is available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Bladder Cancer
  Interventions: Diagnostic Test: Functional drug screen
- Kidney Cancer
  Interventions: Diagnostic Test: Functional drug screen
- Melanoma
  Interventions: Diagnostic Test: Functional drug screen
- Sarcoma
  Interventions: Diagnostic Test: Functional drug screen
- Glioblastoma
  Interventions: Diagnostic Test: Functional drug screen
- Head and Neck Cancer
  Interventions: Diagnostic Test: Functional drug screen

INTERVENTIONS:
Diagnostic Test: Functional drug screen — High-throughput ex-vivo drug screen of cells processed directly from solid tumours to determine sensitivity / resistance profiles

SUMMARY:
EVIDENT's aim is to test if ex vivo drug screening can predict whether patients with solid cancers will respond, or not respond, to standard care treatments. Patients undergoing standard care surgery to excise their tumour, those undergoing a biopsy, or those having a fluid aspirate of a solid tumour with surplus tissue available after diagnostic use will be eligible for this study. The specimen will then be assessed with ex vivo drug screening utilising all standard therapies and therapies that are more novel and in early stages of development. The results of the ex vivo drug screen will be compared to the cancer's actual response to standard care treatments for those that undergo therapy to determine how effective the test is at predicting treatment response.

DETAILED DESCRIPTION:
The EVIDENT study is a feasibility / proof of concept study which is designed to determine if ex vivo screening of a patient's solid tumour can predict the effectiveness of standard cytotoxic chemotherapies and targeted inhibitors in solid cancers prior to the patients treatment. We aim to recruit 100 patient to each group starting with the six currently listed, but leave scope to add new groups of different solid cancers in the future.

EVIDENT aims:

* Demonstrate the feasibility of collecting fresh tumour samples within the NHS from patients with solid tumours for ex vivo screening
* Demonstrate that tumour response to drug exposure can be measured and quantified within an ex vivo screening platform
* Collect the participants' clinical outcome data (tumour response and progression free survival) to their standard of care treatment regimes and correlate with results from the ex vivo drug screen
* Identify novel effective therapies
* Investigate the tumour biopsies derived omics to determine the strength of well-established, less well-established biomarkers, and to identify novel biomarkers through correlation with the ex vivo drug screen results

ELIGIBILITY:
Inclusion Criteria:

>16 years of age with a diagnosis of known or suspected solid cancer who will undergo surgery, biopsy, aspirate, or TURBT

Willing to donate a section fresh tumour tissue from surgery, a TURBT, fluid aspirate, or biopsy surplus to diagnostic use

Willing to donate a 9ml blood sample

Able to give written informed consent

Previously treated patients are eligible if:

* Present with a recurrence of a previously treated tumour. This may be a local or metastatic recurrence
* Have undergone treatment for their cancer, but fail to respond to this and progress
* Have received neoadjuvant therapy for their tumour
* Have undergone chemotherapy, targeted therapy, immunotherapy, hormone therapy and or radiotherapy for a previous tumour

Exclusion Criteria:

Patients with a known diagnosis of a blood borne virus (Hepatitis B, Hepatitis C, HIV). (The laboratories where experiments will be conducted do not have the safety facilities to use material containing these pathogens)

Patients with a current positive COVID-19 infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who fit the eligibility criteria who are currently under the care of Sheffield Teaching Hospitals NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Functional drug screen | 6 years
  Collect and functionally screen solid tumours to determine if ex-vivo drug screening can predict effectiveness of standard cytotoxic chemotherapies and targeted inhibitors in solid cancers by correlating ex-vivo results with patients actual response to standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Danson, PhD, FRCP, Principal Investigator — University of Sheffield, Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No